CLINICAL TRIAL: NCT06239571
Title: Resilient Families: A Dyadic Resiliency Intervention for Parents of Babies in the NICU
Brief Title: Resilient Families Open Pilot: Dyadic Resiliency Intervention
Acronym: R-FAM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Victoria A. Grunberg, PhD, Clinical Psychologist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024P000169
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-05

CONDITIONS: Parents
Keywords: Neonatal Intensive Care Unit; Parental mental health; Parental relationships

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dyadic Resiliency Intervention (Experimental): All participants will receive the intervention, a brief dyadic resiliency intervention
  Interventions: Behavioral: Resilient Families (R-FAM)

INTERVENTIONS:
Behavioral: Resilient Families (R-FAM) — Dyadic, resiliency intervention that aims to reduce depression, anxiety, and posttraumatic stress among parents of babies in the NICU

SUMMARY:
The goal is to develop, refine, and test the feasibility and acceptability of a dyadic, resiliency intervention ("Resilient Families;" R-FAM) that aims to reduce emotional distress and improve relationships among parents in the Neonatal Intensive Care Unit (NICU). To achieve this goal, my aims are three-fold: (1) develop R-FAM using stakeholder input from interviews with parent dyads and focus groups with NICU staff; (2) optimize R-FAM through an open pilot with pre/post assessments and exit interviews; and (3) test R-FAM for feasibility and acceptability through a randomized clinical trial of R-FAM compared with a minimally enhanced usual control (MEUC).

DETAILED DESCRIPTION:
The investigators aim to conduct an open pilot trial of the R-FAM program (Resilient Families) with NICU parents (up to N = 6 dyads) followed by an optional brief exit interview. The investigators will determine if the feasibility, acceptability, and fidelity of the program meet a priori benchmarks. The investigators also hope to establish preliminary efficacy that the program reduces parental emotional distress and other study outcomes described in sections below. The investigators will use qualitative data to optimize the intervention and study procedures for future trials.

This Open Pilot trial will include 6 sessions with a clinical psychologist. The intervention will aim to improve coping skills, communication, and stress management. Participants will learn evidence-based skills (e.g., mindfulness, dialectics, problem-solving) to reduce risk for emotional distress.

The primary outcomes for the open pilot will be the feasibility, acceptability, and fidelity of the R-FAM program. Preliminary effectiveness outcomes will also be examined, as in primary and secondary targets and exploratory outcomes (e.g., emotional distress, couple satisfaction, and family impact).

ELIGIBILITY:
Inclusion Criteria:

* Adult parent/legal guardian (and/or their partner) of a baby admitted to the NICU within past week (age ≥ 18)
* Currently in an intimate relationship and will live with baby after NICU discharge
* At least one dyad member is emotionally distressed (HADS >7 on depression or anxiety subscale)
* English fluency/literacy
* Ability and willingness to participate via live video

Exclusion Criteria:

* Baby is expected to pass away (as determined by medical team)
* Current, untreated psychosis or substance dependence/abuse
* Current self-report of suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Depression | Baseline to end of intervention (6 weeks)
  Level of depression endorsed on Hospital Anxiety & Depression Scale and Edinburgh Postnatal Depression Scale, from 0-30 with 30 indicating highest depression
Anxiety | Baseline to end of intervention (6 weeks)
  Level of anxiety endorsed on Hospital Anxiety & Depression Scale, from 0-21 with 21 indicating highest anxiety
Posttraumatic Stress | Baseline to end of intervention (6 weeks)
  Level of posttraumatic stress endorsed on Impact of Event Scale-6, from 6-24 with 24 indicating highest posttraumatic stress

SECONDARY OUTCOMES:
Couple relationship functioning | Baseline to end of intervention (6 weeks)
  Couple satisfaction as reported on Couple Satisfaction Index, from 0-21 with 21 indicating highest couple satisfaction
Family Impact | Baseline to end of intervention (6 weeks)
  Impact of child's illness as reported on Family Impact Scale, Revised, from 0-75 with 75 indicating lowest impact on family

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Grunberg, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mass General Brigham, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No